CLINICAL TRIAL: NCT01228214
Title: Randomized Double-Blind Placebo-Controlled Study of Pyrazinoylguanidine Hydrochloride (Amiloride) in Subjects With Coronary Artery Disease
Brief Title: Novel Treatment for Coronary Artery Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Carabobo (Other)
Collaborators: Clinical Research Unit at the Instituto Docente de Urologia (Unknown); Northern Metropolitan Hospital (Unknown); Venezuelan Foundation of Heart Failure (Other)
Responsible Party: Principal Investigator, Antonio Delgado Leon, MD, Prof. of Medicine, MD, University of Carabobo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIC-3 2007
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nitrates; Clopidogrel; Aspirin; Amiloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amiloride,nitrates,clopidogrel,aspirin (Experimental): Comparative Efficacious Research
  Interventions: Drug: amiloride
- Placebo,nitrates,clopidogrel,aspirin (Placebo Comparator): Comparative Efficacious Research
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo 5mg/daily for 12 months
  Other Names: nitrates (40mg/daily for 12 months); clopidogrel(75mg/daily for 12 months); aspirin (80mg/daily for 12 months)
  Arms: Placebo,nitrates,clopidogrel,aspirin
Drug: amiloride — 5mg/daily for 12 months
  Other Names: nitrates (40mg/daily for 12 months); clopidogrel(75mg/daily for 12 months); aspirin (80mg/daily for 12 months)
  Arms: Amiloride,nitrates,clopidogrel,aspirin

SUMMARY:
Treatment of coronary artery disease is a major health care problem across the entire word, and the United States. Unfortunately, despite a number of medical advances, diagnostic procedure, or epidemiological studies, the treatment of these patients remain complex, and and at times frustrating. In fact, the COURAGE trial conducted in 50 centers across United States and Canada documented that drug treatment, coronary interventions or both were not effective solution in coronary artery diseases.

A novel approach has recently been developed, based on the critical role of the potassium (K) content in red-blood-cell in myocardial oxygenation, since oxygen and K binding by hemoglobin (red-blood-cell) occurs simultaneously in blood passing through the lungs, whereas in the organs as the heart, the hemoglobin release both Oxygen and K ions.

This apparently simple mechanisms occurs in human blood in all individuals but could be altered in subjects with acquired or hereditable defect in red-blood-cell K content, as in hypertensives or CAD patients.

DETAILED DESCRIPTION:
Treatment of Cardiovascular Diseases (CVD) is a major health care problem across the entire word, and particularly in the United States. In fact, these life-threatening disorders are a major cause of emergency medical care and hospitalization in the United States, and according the National Center for Health Statistics (NCHS) there were approximately 1,565,000 hospitalizations for primary or secondary diagnosis of an acute coronary syndrome (ACS), 669,000 for unstable angina (UA) and 896,000 for myocardial infarction (MI). In the 2003, NCHS reported 4,497,000 visits to emergency departments for primary diagnosis of CVD, wherein the average age of a person having a first heart attack is calculated at 65.8 years for men and 70.4 years for women.

Further studies provided by the Heart Disease and Stroke Statistics-2007 Update, of the American Heart Association, reported an estimated 79 400 000 American adults (1 in 3) have 1 or more types of CVD. Of these, and 37 500 000 are estimated to be age 65 or older. As a separate diagnosis, high blood pressure or hypertension, accounts for approximately 72 000 000 of patients (defined as systolic pressure 140 mm Hg or greater and/or diastolic pressure 90 mm Hg or greater, taking antihypertensive medication), coronary heart disease (CHD) for approximately 15 800 000 patients, myocardial infarction for approximately 7 900 000 patients, and angina pectoris (chest pain secondary to ischemic heart disease) for approximately 8 900 000 patients.

Although the treatment of angina (chest pain secondary to ischemic heart disease and one of the most common and early symptom of coronary artery disease) can be tracked as far as 1880's, it still represents a medically unresolved problem. Indeed, treatment of angina in particular, as well as associated condition as ACS, UA, and MI, involves a large number of life-style change recommendations, dietetic advice, drugs, coronary artery intervention, or coronary bypass surgery aimed to improve symptoms, quality of life of patients, and even primary or secondary prevention of the CVD. Unfortunately, despite a century of medical advances and epidemiological studies, the current approach to CVD, and coronary artery disease remain complex, and at times frustrating.

Among some of the proposals to combat CVD, have included the single "polypill"(aspirin + statin + 3 blood pressure lowering agents in half dose, and folic acid) as a strategy to reduce CVD by more than 80% remains presently unresolved, regression of coronary atherosclerosis by using Simvastatin and intravascular ultrasound study was determined to be unpractical. It remains to be determined whether these changes will translate to meaningful reductions in clinical events, or whether new antithrombotic agents for these CVD patients can provide an adequate solution. However, the overarching determination in view of the purported successes to date remains whether these results in highly selected patient populations can be matched to the real-world treatment of acute coronary syndromes.

In a recent study called the COURAGE Trial (Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation) conducted in 50 hospital centers across the United States and Canada showed that optimal drug treatment with percutaneous coronary interventions (PCI) for stable coronary artery disease, was not more effective than optimal medical therapy alone for preventing cardiovascular events, hospitalization or death, suggesting that drugs, surgical procedures or both were not a statistically effective solution for CHD.

For more than a century, hemodynamic mechanisms involving the coupled tissue O2/CO2 gas exchange and ion H/K transport by Hemoglobin (Hb) in red blood cells (RBC) have been well known to the scientific community, and has been termed the so-called Bohr/Haldane Effect. Data to date has been shown that the RBC has a number of critical roles in maintaining normal vascular function, blood flow, tissue oxygenation and acid-base regulation. These critical roles, including the nitric oxygen (NO) transport, NO synthetase expression, platelet aggregation, vascular rheology, and endothelial function, have been the subject of extensive studies by many investigators. Unfortunately, and despite such multiple integrated functions to maintain tissue oxygenation in health and diseases states, the role of RBC has never been of interest in the therapeutic approach of patients with CHD, specially the ischemic condition of ACS, UA or MI.

In this context, the evidence from our laboratory that erythrocytes have a critical role in body K homeostasis, along with the finding of a hereditable defect in erythrocyte K uptake in hypertensives, and 46% of their normotensive (adolescents, young adults) offspring, led us to assess whether a defective K uptake could impair the regulation of H/K exchange and oxygen delivery in CAD. Since then, a Patent Application whose filed in the USPTO,and a simple medical device for intracellular K measurement in red blood cell by miniature K and Na ion-selective electrode was proposed in conjunction with the University of Michigan.

Although many drugs were tested in order to improve or correct the defective red cell K transport, the most promising compound was the 3,5-diamino-6-chloro-N- [diaminomethylene]pyrazinecarboxamide dihydrate derivative, amiloride hydrochloride recently published as a new drug patent application.

The drug originally tested in hypertensives with low RBC K uptake, independently of cell Na content, dietary intake or drugs, became an effective and predictable method to improve RBC K homeostasis that is critically related to other red-cell functions, such as the pH regulation and oxygen delivery. More important, the observation that reversal of the abnormal RBC K content was associated with a decline and better control of BP, fasting plasma glucose, and regression of ST-T alteration related to LVH or CHD, led us to evaluate the role of RBC in the mechanism of H/K exchange, tissue oxygenation in health and disease states.

This Clinical Trial will address the effects of Amiloride in RBC K uptake, and consequently the simultaneous tissue H/K and O2/CO2 exchange, its therapeutic effect on BP control and possible improvement on Angina, Duke Treadmill Score, and ST-T alteration of LVH or CAD.

METHODS OF TREATMENT

Each patient will be prospectively evaluated in order to assess the effects of Amiloride on reversion of angina and ECG alterations of ischemia in CAD. After written consent, the subject will enter the Double-Blind trial of Amiloride Vs Placebo along whit the optimal treatment for Angina and CHD. Amiloride (5 to 10 mg) will be given daily, before breakfast, while other medication for angina, and associated diseases as hypertension or diabetes, were continued. Each patient will be clinically evaluated for angina, dyspnea, or arrhythmias at 1-week, 1, 3, 6 months period. Serial ECG, Ion Transport Studies, BIA, non-invasive hemodynamic and clinical biochemistry will be obtained at 1, 3, 6 months follow-up period. Echocardiograms were obtained basal and 6- months period. In this trial, each subject with plasma ionized calcium (≤1.0 mmol/l) will received 1g of Ca- gluconolactate until the level was ≥1.0 mmol/l.

Following the first 3-month trial, patients with reversion of angina and improvement of ECG abnormalities of ischemia will have low doses of amiloride (5 to 7.5 mg), while nitrates, B-blockers or Calcium Channel Blockers will be progressively discontinued, if no evidence of angina occurred, and if no new no ECG ST-T alteration of ischemia developed. Therefore, amiloride with/without aspirin, Statins and medication for hypertension or diabetes, will be the established treatment until the end of trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 35-75 years having angina (Canada Cardiovascular Society Class II-IV)
2. Essential Hypertension defined as taking at least 1 anti-hypertensive medication, or average systolic blood pressure ≥140 mm Hg, or diastolic blood pressure ≥90 mmHg
3. ST-T changes of LVH (Romhilt-Estes or Framingham Heart Study criteria, with typical LV strain pattern, or isoelectric, inverted or biphasic T waves)
4. ST-T changes of ischemia in resting ECG (ST depression, isoelectric, biphasic, negative or inverted T-waves)
5. Serum potassium < 5.0 mmol/L prior to randomization
6. Negative pregnancy test in child-bearing potential women
7. Willing to comply with scheduled visits
8. Informed consent form signed by the subject

Exclusion Criteria:

1. Resistance hypertension despite 3-drugs treatment
2. Myocardial infarction in past 90 days
3. Coronary artery bypass graft surgery in past 90 days
4. Atrial fibrillation with a resting heart rate > 90 bpm
5. Percutaneous coronary intervention in past 30 days
6. Implanted Pacemaker
7. Stroke in past 90 days
8. Left or Right Ventricular Branch Block
9. Aldosterone antagonist or K sparing drug in last 7 days
10. Intolerance to amiloride
11. Lithium use
12. Current participation in any other therapeutic trial
13. Any condition that may prevent the subject from adhering to the trial protocol
14. History of hyperkalemia (K ≥5.5 mmol/L) in the past six months or K >5.0 mmol/L within 2 weeks
15. Chronic renal dysfunction
16. Liver disease
17. Chronic pulmonary disease
18. Significant uncorrected valvular heart disease

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Regression of Angina Without Recurrence | Baseline, 1, 3, 6 and 12 Months during the first year trial, and every 6-months in the 2nd year period
  Evaluation of Angina Class according the Canadian Society of Cardiology (CCS)
Regression of ST-T and T-waves Alterations of Myocardial Ischemia | Baseline, 1, 3, 6 and 12 Months during the first year trial, and every 6-months in the 2nd year period
  Evaluation according the Minnesota Code
RBC Potassium Content | Baseline, 1, 3, 6 and 12 Months during the first year trial, and every 6-months in the 2nd year period
  Obtained by a novel accurate method developed in our laboratory (Nutr Metab Cardiovasc Dis. 2002 Jun;12(3):112-116

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Delgado-Leon, MD, Study Chair — University of Carabobo; Carlos L Delgado-Leon, MD, Study Director — Venezuelan Foundation of Heart Failure; Antonio R Delgado-Almeida, MD, FAHA, FACC, APS, Principal Investigator — Clinical Research Unit at Docent Institute of Urology
Locations (1):
- Hypertension Research Unit, Valencia, Carabobo, Venezuela

REFERENCES:
- [Background] Delgado-Almeida A. Assessing cell K physiology in hypertensive patients. A new clinical and methodologic approach. Am J Hypertens. 2006 Apr;19(4):432-6. doi: 10.1016/j.amjhyper.2005.09.013. PMID 16580582
- [Background] Delgado MC, Delgado-Almeida A. Red blood cell K+ could be a marker of K+ changes in other cells involved in blood pressure regulation. J Hum Hypertens. 2003 May;17(5):313-8. doi: 10.1038/sj.jhh.1001527. PMID 12756403
- [Background] Delgado-Almeida A. Unexpected therapeutic response to spironolactone: a prospective debate on aldosterone and potassium ion in hypertension. Hypertension. 2007 Nov;50(5):e164-5; author reply e166. doi: 10.1161/HYPERTENSIONAHA.107.099408. Epub 2007 Sep 10. No abstract available. PMID 17846345
- [Background] Delgado-Almeida A. Reinterpreting sodium-potassium data in salt-sensitivity hypertension: a prospective debate. Hypertension. 2005 Feb;45(2):e4; author reply e4. doi: 10.1161/01.HYP.0000154194.49725.b7. No abstract available. PMID 15630043
- [Background] Delgado-Almeida A. Critical value of the electrocardiogram in LVH: from predictive index to therapeutic reassessment. Hypertension. 2005 Feb;45(2):e6; author reply e6. doi: 10.1161/01.HYP.0000151782.93734.de. No abstract available. PMID 15583072
- [Background] Delgado MC, Delgado-Almeida A. Red blood cell potassium and blood pressure in adolescents: a mixture analysis. Nutr Metab Cardiovasc Dis. 2002 Jun;12(3):112-6. PMID 12325467
- [Background] Delgado MC, Delgado-Almeida A. Abnormal Potassium. In: Mohler III ER, Townsend RR (eds). Advanced Therapy in Hypertension and Vascular Disease. BC Decker Inc. Publisher, Ontario, Canada. 2006:291-296.
- [Background] Weder AB, Delgado MC, Zhu X, Gleiberman L, Kan D, Chakravarti A. Erythrocyte sodium-lithium countertransport and blood pressure: a genome-wide linkage study. Hypertension. 2003 Mar;41(3 Pt 2):842-6. doi: 10.1161/01.HYP.0000048703.16933.6D. Epub 2002 Dec 23. PMID 12624006
- [Background] Delgado MC. Potassium in hypertension. Curr Hypertens Rep. 2004 Feb;6(1):31-5. doi: 10.1007/s11906-004-0008-6. PMID 14972087